CLINICAL TRIAL: NCT06185803
Title: Predictors of Anterior Patellofemoral Pain After Anterior Cruciate Ligament Reconstruction.
Acronym: SPEDAL
Status: Active, not recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Vivactis M2Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-12-026
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: anterior cruciate ligament reconstruction — anterior cruciate ligament reconstruction

SUMMARY:
Observational, ambispective, longitudinal, monocentric, open cohort study of a population of adult patients operated on for ACL reconstruction and receiving postoperative follow-up.

DETAILED DESCRIPTION:
On a large population of adult patients operated on for anterior cruciate ligament reconstruction and followed over a 12-month period under standard medical practice conditions.

Primary objective: to investigate, six months after surgery, the presence of patellofemoral pain and to evaluate the factors predictive of the occurrence of such pain.

Secondary objectives:

* Evaluate the incidence of patellofemoral pain at 12 months.
* Compare the functional status of patients with and without patellofemoral pain at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient who has been informed of the research and does not object to data collection
* Patient who has undergone or is about to undergo ACL ligamentoplasty surgery
* Regularly followed-up patient for whom the data required by the protocol will be available in the medical record History of contralateral ACL rupture

Exclusion Criteria:

* History of associated fracture
* History of multi-ligament reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion population will be described according to all patient characteristics.
  Quantitative variables will be described by their number, mean, standard deviation, median, extreme values and missing data. Qualitative variables will be described by their number, percentage and missing data. Bilateral 95% confidence intervals will be provided if the criterion is considered relevant.
  The population will be described overall and in each group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Anterior patellofemoral pain | Month 6
  The presence of anterior patellofemoral pain at 6 months post-op was the primary endpoint of the study.

SECONDARY OUTCOMES:
Returning to sport | Month 6
  Returning to sport after anterior cruciate ligament (ACL) reconstruction requires optimal physical and psychological recovery. The Anterior Cruciate Ligament-Return-to-Sport after Injury (ACL-RSI) scale is the first tool to assess this psychological dimension.
  It consists of 12 questions with answers rated from 0 to 10 on a simple numerical scale
Returning to sport | Month 12
  Returning to sport after anterior cruciate ligament (ACL) reconstruction requires optimal physical and psychological recovery. The Anterior Cruciate Ligament-Return-to-Sport after Injury (ACL-RSI) scale is the first tool to assess this psychological dimension.
  It consists of 12 questions with answers rated from 0 to 10 on a simple numerical scale
Subjective knee assessment | Month 6
  The International Knee Documentation Committee Subjective Knee Form is a self-administered questionnaire divided into three sections (symptoms, sports activities, function).
  Its score ranges from 0 (worst situation) to 100 (no restrictions on daily activities and sports, and no symptoms).
Subjective knee assessment | Month 12
  The International Knee Documentation Committee Subjective Knee Form is a self-administered questionnaire divided into three sections (symptoms, sports activities, function).
  Its score ranges from 0 (worst situation) to 100 (no restrictions on daily activities and sports, and no symptoms).
Subjective symptoms assessment | Month 6
  The Kujala Anterior Knee Pain Scale (Kujala AKPS) is a questionnaire used to assess subjective symptoms such as functional limitations and anterior knee pain. It comprises 13 items: 6 concerning the patient's activities (walking, running, jumping, stairs, squatting, prolonged sitting), 7 concerning the patient's symptoms (lameness, unloading, swelling, maltracking of the patella, muscle atrophy, flexion deficit).
  The score ranges from 0 (highly symptomatic patient) to 100 (asymptomatic patient). Patients with a score of 70 are considered to have moderate disability.
Subjective symptoms assessment | Month 12
  The Kujala Anterior Knee Pain Scale (Kujala AKPS) is a questionnaire used to assess subjective symptoms such as functional limitations and anterior knee pain. It comprises 13 items: 6 concerning the patient's activities (walking, running, jumping, stairs, squatting, prolonged sitting), 7 concerning the patient's symptoms (lameness, unloading, swelling, maltracking of the patella, muscle atrophy, flexion deficit).
  The score ranges from 0 (highly symptomatic patient) to 100 (asymptomatic patient). Patients with a score of 70 are considered to have moderate disability.
Sporting and occupational physical activity assessment | Month 6
  The Tegner activity-level scale is a scale of sporting and occupational physical activity: from 0 (occupational disability due to knee) to 10 (competitive sport such as soccer or rugby at national or international level).
  The scale was originally developed to measure activity following knee injuries, and validated for monitoring ACL ruptures following ligamentoplasty.
Sporting and occupational physical activity assessment | Month 12
  The Tegner activity-level scale is a scale of sporting and occupational physical activity: from 0 (occupational disability due to knee) to 10 (competitive sport such as soccer or rugby at national or international level).
  The scale was originally developed to measure activity following knee injuries, and validated for monitoring ACL ruptures following ligamentoplasty.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No